CLINICAL TRIAL: NCT05878171
Title: Preference of Life-Sustaining Treatment Among Patients With End Stage Renal Disease
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 202303044RINC
Record Dates: First submitted 2023-05-07; First posted 2023-05-26 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: End Stage Renal Disease
Keywords: Life-Sustaining Treatment,End Stage Renal Disease,Preference
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although patients with kidney disease can rely on dialysis to prolong their lives, the complexity of the disease, the variability of the course of the disease, and the uncertainty of the prognosis often delay the discussion of issues at the end of life, and the deterioration of the condition often makes it impossible for the patient to express clearly or rationally. Treatment thoughts or preferences. Sufficient time is needed to think and discuss issues related to life treatment. Discuss with patients as soon as possible to help draw up end-of-life care plans, help patients realize end-of-life care preferences, assist family members to make complex treatment decisions, and alleviate medical providers' moral distress. Domestic life-sustaining treatment research is mostly signed by DNR for cancer patients and retrospective investigation of medical records, and seldom focuses on kidney disease patients and life-sustaining treatment survey preferences other than DNR content. This study sought to understand patients with kidney disease's preferences for life-sustaining care during disease progression, and to understand whether prognostic perceptions, symptom distress, dementia, and decision conflict affect patients' preferences. Pre-collected convenient sampling is expected to include 200 patients diagnosed with chronic kidney disease stage 5 or end-stage renal disease, including patients who have received regular dialysis. The survey will be conducted with a single questionnaire. There are five questionnaires, including: demographic characteristics, chronic kidney disease prognosis cognition And life-support treatment information questionnaire, short-form recall symptom assessment scale, loss of memory scale and decision-making conflict scale; after the researcher explains, the patient fills in by himself or the researcher fills in after the patient answers. It is expected that the results of the study will help clinical practitioners to understand the changes in the management of medical care for kidney disease patients when the disease worsens and assist in the management of patients' medical care, echoing the importance of advancing medical care planning in this population, for the future development of kidney disease A reference for care guidelines for debilitated patients, thereby improving care quality and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 years old.
2. Patients diagnosed with chronic kidney disease stage V or end-stage renal disease, and glomerular filtration rate less than 15ml/min/1.73m2; or patients receiving regular blood or peritoneal dialysis treatment.
3. Those who have normal cognitive function (such as: able to read newspapers and magazines, and communicate with others), and can communicate in Mandarin and Taiwanese.

Exclusion Criteria:

1. Severe cognitive impairment or visual or hearing impairment that makes it impossible to answer questions.
2. Critically ill patients.
3. Patients with chronic mental illness or their related diagnosis records.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic kidney disease stage V or end-stage renal disease, and glomerular filtration rate less than 15ml/min/1.73m2; or patients receiving regular blood or peritoneal dialysis treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Preference for end-of-life life-sustaining treatment for patients with end-stage renal disease | one year
  This study aimed to investigate end-stage renal disease treatment and end-of-life life-sustaining treatment preferences in patients with renal failure. Life-sustaining treatment preferences include cardiac resuscitation, endotracheal intubation, mechanical ventilation, blood transfusion, antibiotics, and artificial nutrition and fluids. And life support treatment preference is divided into three aspects: preference choice, clear understanding, and certainty for preference data investigation: (1) For each life support treatment preference choice, "absolutely", "maybe", "may not" " Never"; (2) Are you aware of your preferences for each life-sustaining treatment clearly enough to select a "yes" and "no" option; (3) Are you confident in choosing each life-sustaining treatment? "Yes" and "No" options.
The influencing factors of life-sustaining treatment preference in patients with end-stage renal disease | one year
  The life-sustaining treatment that patients with ESRD are willing to receive at the end of life will be affected by demographic characteristics, that is, collecting patients' sex, age, time of kidney disease diagnosis, frequency of dialysis, religion, occupational status and laboratory reports; prognostic perception will ask patients Self-prognosis expectations are less than 5 years, 5 to 10 years, greater than 10 years and uncertain; MSAS-SF is used to investigate the symptoms of patients within a week, and can also be compared with cancer and other diseases; Demoralization Scale-Mandarin Version is used to describe the degree of pain in the past two weeks, describe the pain of the patient, judge the severity of the patient's low morale, predict suicidal behavior, evaluate the quality of life and screen the diagnosis of depression but face survival crisis and lose the meaning of life of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Shiuan Kuo, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taipei University of Nursing and Health Sciences, Taipei

IPD SHARING:
Plan to Share IPD: Yes
height and weight,BUN,Cre,eGFR, pH,HCO3,CO2,HB,WBC,Plt,CRP,Na,K,Ca,P,Alb,HBA1c,Cardiac ultrasound,Cardiac Catheterization,computed tomography
Supporting Information: ICF
Time Frame: starting 2 months after publication
Access Criteria: File and encode the data through Microsoft Excel conversion, and use SPSS 22.0 software for data analysis.
  Descriptive statistics describe the distribution of data, and inferential statistics set a 95% confidence interval, and a p value less than 0.05 is considered significant. Chi-square test (Chi-square) and ANOVA were used to detect whether the patient's preference for life-sustaining treatment was related to the basic demographic status, dialysis treatment situation, prognosis cognition, symptom distress and dementia. Age, duration of renal disease, ADL, frequency of cardiopulmonary resuscitation and chance of self-conscious disease recovery were tested by independent sample t test. Pearson's product-difference correlation coefficient describes the relationship between each variable and life-sustaining treatment preference, and logistic regression predicts important factors that affect patients' life-sustaining treatment preference.

REFERENCES:
- [Background] Saeed F, Sardar M, Rasheed K, Naseer R, Epstein RM, Davison SN, Mujtaba M, Fiscella KA. Dialysis Decision Making and Preferences for End-of-Life Care: Perspectives of Pakistani Patients Receiving Maintenance Dialysis. J Pain Symptom Manage. 2020 Aug;60(2):336-345. doi: 10.1016/j.jpainsymman.2020.03.009. Epub 2020 Mar 20. PMID 32201311
- [Result] O'Hare AM, Kurella Tamura M, Lavallee DC, Vig EK, Taylor JS, Hall YN, Katz R, Curtis JR, Engelberg RA. Assessment of Self-reported Prognostic Expectations of People Undergoing Dialysis: United States Renal Data System Study of Treatment Preferences (USTATE). JAMA Intern Med. 2019 Oct 1;179(10):1325-1333. doi: 10.1001/jamainternmed.2019.2879. PMID 31282920
- [Result] Bernacki GM, Engelberg RA, Curtis JR, Kurella Tamura M, Brumback LC, Lavallee DC, Vig EK, O'Hare AM. Cardiopulmonary Resuscitation Preferences of People Receiving Dialysis. JAMA Netw Open. 2020 Aug 3;3(8):e2010398. doi: 10.1001/jamanetworkopen.2020.10398. PMID 32833017
- [Result] Saeed F, Sardar MA, Davison SN, Murad H, Duberstein PR, Quill TE. Patients' perspectives on dialysis decision-making and end-of-life care . Clin Nephrol. 2019 May;91(5):294-300. doi: 10.5414/CN109608. PMID 30663974
- [Result] Scherer JS, Milazzo KC, Hebert PL, Engelberg RA, Lavallee DC, Vig EK, Kurella Tamura M, Roberts G, Curtis JR, O'Hare AM. Association Between Self-reported Importance of Religious or Spiritual Beliefs and End-of-Life Care Preferences Among People Receiving Dialysis. JAMA Netw Open. 2021 Aug 2;4(8):e2119355. doi: 10.1001/jamanetworkopen.2021.19355. PMID 34347059